CLINICAL TRIAL: NCT01787019
Title: Initiation of Oral Feeding at 30 Versus 33 Weeks Postmenstrual Age
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Health Science Center, Houston (Other)
Responsible Party: Principal Investigator, Kathleen Kennedy, Professor of Pediatrics, The University of Texas Health Science Center, Houston
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Age of Oral Feeding
Record Dates: First submitted 2013-02-04; First posted 2013-02-08 (Estimated); Last update posted 2016-05-13 (Estimated); Status verified 2016-05

CONDITIONS: Prematurity
MeSH Terms: conditions — Premature Birth

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- 30 weeks (Experimental): initiation of oral feedings at 30 weeks
  Interventions: Other: Oral feeding
- 33 weeks (Active Comparator): initiation of oral feedings at 33 weeks
  Interventions: Other: Oral feeding

INTERVENTIONS:
Other: Oral feeding

SUMMARY:
The purpose of the study is to determine if earlier initiation of oral (by mouth as opposed to tube) feedings in premature infants results in earlier attainment of full oral feedings and/or discharge.

DETAILED DESCRIPTION:
Infants will be enrolled and randomized at 30 0/7 weeks postmenstrual age. The Earlier Oral Feeding group will initiate oral feedings at 30 0/7 weeks postmenstrual age. The Later Oral Feeding group will initiate oral feedings at 33 0/7 weeks postmenstrual age. The number of oral feeding attempts will be advanced according to a feeding progression protocol for both groups. Successful completion of a feeding is defined as oral completion of the full volume of a feeding within 30 minutes, without a bradycardic episode (heart rate <100 beats per minute) or desaturation (oxygen saturation decrease >5% from baseline values). If infant does not successfully complete >95% of the total prescribed volume of a feeding, the remainder of the volume will be supplied via gastric tube. All oral feedings will be performed by bedside nurses, or by a parent with observation by the nursing staff, with continuous cardiorespiratory and pulse oximetry monitoring. Individual oral feeding attempts for both groups will continue until one of the following occurs despite appropriate pacing of the feeding: 1) the feeding is completed 2) feeding duration of 30 minutes 3) adverse event during a feeding [multiple bradycardic episodes (3 episodes of heart rate <100 beats per minute), bradycardia with choking episode, single severe bradycardia (heart rate <60)]. If the infant experiences an adverse event during an oral feeding attempt, oral feeding attempts will be held for 2 days.

ELIGIBILITY:
Inclusion Criteria:

* Gestational age <= 29 weeks at birth
* Tolerating enteral feedings for at least 3 days before 30 weeks postmenstrual age

Exclusion Criteria:

* Neurologic, cardiac, respiratory, or gastrointestinal disorders that interfere with oral feeding

Max Age: 7 Weeks | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 66 (Actual)
Dates: Start 2013-01; Primary Completion 2016-04 (Actual); Study Completion 2016-04 (Actual)

PRIMARY OUTCOMES:
Postmenstrual age at full oral feeding | until hospital discharge (typically 36 weeks postmenstrual age)
  defined as the infant orally consuming the volume of formula/breastmilk as prescribed by the attending physician without requiring gavage feedings for 2 days

SECONDARY OUTCOMES:
postmenstrual age at discharge | until hospital discharge (typically 36 weeks postmenstrual age)
growth between enrollment and 36 weeks postmenstrual age | until hospital discharge (typically 36 weeks postmenstrual age)

OTHER OUTCOMES:
average FiO2 | at 33 weeks postmenstrual age
use of positive pressure (yes/no) | 33 weeks postmenstrual age

CONTACTS AND LOCATIONS:
Locations (1):
- Children's Memorial Hermann Hospital, Houston, Texas, United States